CLINICAL TRIAL: NCT07353138
Title: The Relationship Between Preoperative Neutrophil-to-Lymphocyte Ratio and Hemogram Parameters and Early Postoperative Pain Scores in Patients Undergoing Septorhinoplasty
Brief Title: Preoperative Neutrophil-to-Lymphocyte Ratio and Early Postoperative Pain After Septorhinoplasty
Status: Not yet recruiting | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, İlke Dolgun, Assos.Prof., Istinye University
Other Study IDs: 323-2025
Record Dates: First submitted 2026-01-07; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Neutrophil-to-Lymphocyte Ratio; Septorhinoplasty
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational Study — Not applicable. This is a prospective observational study. No intervention or alteration to standard treatment protocols will be performed. Clinical and laboratory data obtained during routine care, including preoperative hemogram parameters and early postoperative pain scores, will be recorded and analyzed without influencing patient management.

SUMMARY:
This prospective, observational study investigates the relationship between early oxygen exposure and oxidative stress in adult intensive care unit patients with sepsis or septic shock. Fraction of inspired oxygen (FiO₂) administered during the first 24 hours of ICU admission will be recorded and analyzed in relation to changes in the uric acid/albumin ratio (UAR), a biomarker reflecting oxidative burden and inflammation. Serum uric acid and albumin levels will be measured at baseline and at 24 hours, and the percentage change in UAR will be calculated. Secondary analyses will examine associations between UAR changes, oxygenation indices, and 28-day mortality. The study aims to determine whether higher FiO₂ exposure is associated with increased oxidative stress and to evaluate the potential role of UAR as a clinically accessible marker of oxygen-related oxidative injury in septic ICU patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18-65 years
* Patients undergoing elective septorhinoplasty
* Surgery performed under general anesthesia
* Complete recording of early postoperative VAS pain scores, Aldrete scores, NUDES scores, and vital signs in the Post-Anesthesia Care Unit (PACU)
* Preoperative complete blood count (hemogram) performed within 30 days prior to surgery
* Clinical records and hospital information system data that are complete, accessible, and adequate for analysis

Exclusion Criteria:

* Patients undergoing emergency surgery
* Septorhinoplasty combined with additional major surgical procedures (e.g., advanced ENT or maxillofacial surgery)
* Presence of known hematological disease, active infection, immunosuppressive therapy, or advanced liver or renal failure
* Chronic opioid use or regular analgesic medication use in the preoperative period
* History of significant clinical events between the preoperative hemogram and surgery that could alter inflammatory status (e.g., infection, hospitalization, additional surgery)
* Incomplete or missing data regarding preoperative hemogram parameters or PACU pain scores

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18-65 years who undergo elective septorhinoplasty under general anesthesia. All participants are managed according to standard clinical practice and are admitted to the Post-Anesthesia Care Unit (PACU) postoperatively, where early pain assessments and routine clinical monitoring are performed. Eligible patients have a complete preoperative hemogram obtained within 30 days prior to surgery and comprehensive postoperative records, including pain scores and vital signs. Patients with conditions or treatments that could significantly affect inflammatory markers or pain perception are excluded to ensure a homogeneous study population
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Early Postoperative Pain Severity | Within the first 60 minutes after admission to the Post-Anesthesia Care Unit (PACU).
  early postoperative pain severity, as measured using the Visual Analog Scale (VAS). 0: no pain, 10 worst pain

REFERENCES:
- [Background] Sachidananda R, Malipatil A, Joshi V, Hosamani A, Haranagatti A, Kurugodiyavar MD. Relationship between neutrophil-lymphocyte ratio and postoperative pain in cesarean section patients done under subarachnoid block: A prospective observational study. J Anaesthesiol Clin Pharmacol. 2025 Jul-Sep;41(3):464-469. doi: 10.4103/joacp.joacp_213_24. Epub 2024 Dec 16. PMID 40635819
- [Background] Yildiz Altun A, Demirel I, Bolat E, Ozcan S, Altun S, Aksu A, Bestas A. The Relationship Between the Preoperative Neutrophil-to-Lymphocyte Ratio and Postoperative Nausea and Vomiting in Patients Undergoing Septorhinoplasty Surgery. Aesthetic Plast Surg. 2019 Jun;43(3):861-865. doi: 10.1007/s00266-019-01325-5. Epub 2019 Feb 14. PMID 30767038